CLINICAL TRIAL: NCT04864990
Title: Dyspnea in Idiopathic Pulmonary Fibrosis (IPF): Multidimensional Assessment and Correlations With Lung Function
Brief Title: Dyspnea and Idiopathic Pulmonary Fibrosis
Acronym: DYS-PID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Santelys Association (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_62; 2020-A00803-36 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Longitudinal prospective exploratory study on the evolution of dyspnea, in its sensory and affective dimensions, in patients followed for idiopathic pulmonary fibrosis (IPF), between inclusion and a 6-month evaluation

DETAILED DESCRIPTION:
Dyspnea is a multidimensional experience involving a sensory component and an affective component. To better understand this symptom in IPF, this study will describe the different component of dyspnea and their evolution between inclusion and a 6-month evaluation in IPF patients.

There is no strong correlation between the intensity of dyspnea and respiratory function impairments. Innovative techniques demonstrated abnormalities in ventilation variability and pulmonary compliance in patients with interstitial lung disease. These abnormalities could be more relevant to explain dyspnea. The objective of this work is also to assess the link between the different dimensions of dyspnea and respiratory functional parameters, ventilation variability and ventilatory mechanics measured by impulse oscillometry technique.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of IPF according to ATS/ERS guidelines
* dyspnea at rest (VAS ≥ 1) or on exertion (mMRC ≥ 1)

Exclusion Criteria:

* diffuse interstitial lung disease other than IPF
* other significant chronic pathology that may cause dyspnea: chronic obstructive pulmonary disease, asthma, heart failure, anemia, obesity (non-exhaustive list), except for pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with a diagnosis of idiopathic pulmonary fibrosis (IPF) and reporting dyspnea
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Evolution of the sensory and affective components of dyspnea | baseline, 6 months
  Description and changes in sensory (SQ) and affective (A2) scores of the Multidimensional Dyspnea Profile (MDP) questionnaire

SECONDARY OUTCOMES:
Evolution of dyspnea during activities of daily living | baseline, 6 months
  Description and changes in San Diego Shortness of Breath Questionnaire (SOBQ) score
Association between the sensory and affective components of dyspnea and quality of life, anxiety symptoms, lung volumes, gas exchanges, ventilation variability, pulmonary compliance, pulmonary hypertension | baseline, 6 months
  Correlation between SQ and A2 scores of the MDP questionnaire and King's Brief Interstitial Lung Disease (K-BILD) questionnaire score, State Trait Anxiety Inventory (STAI-Y2) score, lung volumes measured by plethysmography, DLCO, PaO2, delta of desaturation during the 6-minute walk test, coefficient of variation of the tidal volume at rest, impulse oscillometry reactance, systolic pulmonary artery pressure assessed by cardiac ultrasound
Assess the prevalence of refractory dyspnea | baseline, 6 months
  Description of the prevalence of patients with visual anolog scale at rest > 3 or mMRC scale > 2

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Chenivesse, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Calmette Chu Lille, Lille, France